CLINICAL TRIAL: NCT01693432
Title: A Phase II Study of Docetaxel and S-1 as First-line Chemotherapy in Patients With Advanced Esophageal Cancer
Brief Title: Docetaxel and S-1 for Advanced Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-1202
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Esophageal Neoplasms
Keywords: Esophageal neoplasms; Docetaxel; S-1
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DS (docetaxel+S-1) (Experimental): Treatment will be delivered as a 3-week cycle.
  1. Docetaxel 60 mg/m²IV on day 1
  2. S-1 80 mg/m2/day PO on day 1-14
  Interventions: Drug: DS (docetaxel+S-1)

INTERVENTIONS:
Drug: DS (docetaxel+S-1) — Treatment will be delivered as a 3-week cycle.
  1. Docetaxel 60 mg/m²IV on day 1
  2. S-1 80 mg/m2/day PO on day 1-14
  Other Names: Taxotere; TS-1

SUMMARY:
This study will evaluate the efficacy of docetaxel and S-1 combination chemotherapy in Korean patients with esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer is the ninth most common cancer in male population in Korea. It was estimated that 1,864 new cases of esophageal cancer were reported and 1,434 deaths occurred in Korea in 2005.

Although half of the patients with esophageal cancer initially present with locoregional disease amenable to radical surgery or radiation-based therapy, most patients eventually develop metastatic disease with or without local recurrence.

Chemotherapy plays a major role in palliative therapy and remains to be the primary mode of treatment for the recurrent or metastatic esophageal cancer. Although various chemotherapy regimens are available, esophageal cancer carries a very poor prognosis, with a mean survival time of less than 8.1 months with current chemotherapies used singly or in combination with 5-fluorouracil (5-FU), vindesine, mitomycin, docetaxel, paclitaxel, cisplatin, irinotecan, vinorelbine, or capecitabine. The majority of the trials performed were in small numbers of patients with reported response rates from 15 to 40%.

The response was usually of short duration and there was no survival benefit with single agent chemotherapy. Combination chemotherapy has slightly improved the results in terms of duration of response (3-6 months), but still there was little improvement in overall survival. Therefore, the identification of new active agents is essential to prolong the survival.

Clinical trials of single agent docetaxel have been reported in patients with esophageal cancer and the response rate is about 18-25%.

S-1, a new biochemical modulator of 5-FU, is an oral dihydropyrimidine dehydrogenase(DPD) inhibitory fluoropyrimidine. The advantages of S-1 compared with 5-FU are greater convenience because of its oral formulation and continuous delivery, without intravenous infusion. S-1 is frequently used as a substitute for 5-FU in gastric cancer, but limited data is available for esophageal cancer.

The combination of docetaxel and S-1 is highly active and well tolerated in advanced or recurrent gastric cancer, and the synergistic antitumor activity has been fully elucidated.

Therefore, we will evaluate the efficacy of docetaxel and S-1 combination chemotherapy in Korean patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma or adenocarcinoma of esophagus.
* Unresectable locally advanced, recurrent or metastatic disease.
* Measurable or evaluable disease by RECIST criteria 1.1.
* Minimum age of 18 years.
* ECOG Performance status 0-2.
* Prior chemotherapy is not allowed.
* More than 4 weeks since completion of prior radiotherapy (measurable or evaluable lesions are outside the radiation field)
* Adequate organ functions
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Other tumor type than squamous cell carcinoma and adenocarcinoma
* Previous history of chemotherapy except neoadjuvant or adjuvant chemotherapy without docetaxel and S-1
* Obvious bowel obstruction unrelieved by proper management
* Evidence of serious gastrointestinal bleeding
* Patients with CNS metastases
* Patients with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 6 months, pregnancy, or breast feeding
* Any previous or concurrent malignancy other than non-melanoma skin cancer or in situ cancer of uterine cervix
* Known history of cerebral or leptomeningeal metastases or neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2011-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1.5 years
  Objective response rate will be measured from the rate of complete response (disappearance of disease) and partial response (decrease at least 30% in the sum of the longest diameters of target lesions) by RECIST (response evaluation criteria in solid tumors) guidelines.

SECONDARY OUTCOMES:
Progression free survival | 1.5 years
  Progression free survival time will be measured from the start of study treatment until documented tumor progression, or death due to any cause
Overall survival | 1.5 years
  Overall survival time will be measured from the start of study treatment until death due to any cause
Toxicity profiles | 1.5 years
  adverse events will be descripted and graded using NCI-CTCAE version 4.0
Disease control rate | 1.5 years
  Disease control rate will be measured from the rate of complete response (disappearance of disease), partial response (decrease at least 30% in the sum of the longest diameters of target lesions), and stable disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD) by RECIST (response evaluation criteria in solid tumors) guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Medical Center, Anyang, South Korea

IPD SHARING:
Plan to Share IPD: Undecided